CLINICAL TRIAL: NCT03334643
Title: The Effect of a Dietary Fiber Mix on Glycemic Response in Human: a Pilot Study
Brief Title: Fiber Mix and Glycemic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Liping Zhao PhD, Professor, Professor, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-074m
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Type2 Diabetes Mellitus
Keywords: Type 2 Diabetes; Dietary fiber; Glycemic response
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either the Non-Diabetes or Prediabetes/Diabetes group based on their diagnosis of type 2 diabetes (if any) and their fasting blood glucose concentrations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Diabetes (Experimental): Participants without clinical diagnosis of impaired glucose tolerance or type 2 diabetes and with fasting blood glucose less than 100 mg/dL. They will consume white bread or fiber mix for multiple times over a span of 2 weeks. Changes in blood glucose levels will be monitored.
  Interventions: Dietary Supplement: Fiber mix
- Prediabetes/Diabetes (Experimental): Participants who are clinically diagnosed with impaired glucose tolerance or type 2 diabetes, and those without the above diagnosis but with fasting blood glucose equal to or greater than 100 mg/dL. They will consume white bread or fiber mix for multiple times over a span of 2 weeks. Changes in blood glucose levels will be monitored.
  Interventions: Dietary Supplement: Fiber mix

INTERVENTIONS:
Dietary Supplement: Fiber mix — Participants will test white bread or fiber mix over a span of 2 weeks. During each testing block, each food will be tested twice over two consecutive days. There are 4 testing blocks in total (one for white bread and three for fiber mix).

SUMMARY:
This study determines the acute effect of a dietary fiber mix on blood glucose levels. Participants will consume the fiber mix as a drink and we will monitor changes in blood glucose levels. All participants will consume white bread as the control food.

DETAILED DESCRIPTION:
There is some evidence for increased dietary fiber intake to positively impact on metabolic outcomes in patients with type 2 diabetes, potentially via modulating gut microbial composition and functions. We have developed a dietary fiber mix that is consisted of fiber of various physicochemical properties to maximize the fermentability of the supplement and thus its effects on the gut microbiota. Since the fiber mix also contains nutrients that will raise blood glucose levels, we need to characterize the glycemic response to the fiber mix itself, before we can use it in an upcoming trial to determine the effect of dietary fiber supplementation on the gut microbiota and glycemic control.

Enrolled participants will be assigned to a subject group based on their diagnosis of type 2 diabetes and fasting blood glucose concentrations. Participants who are clinically diagnosed with impaired glucose tolerance or type 2 diabetes will be assigned to the Prediabetes/Diabetes group. For the other participants, those with fasting blood glucose < 100 mg/dL will be assigned to the Non-Diabetes group, and those with fasting blood glucose > 100 mg/dL will be assigned to the Prediabetes/Diabetes group.

Participants will attend 8 food testing visits over 2 weeks. For each visit, participants will attend the research facility in the morning after an overnight fast. They will consume either white bread (with 50 g of available carbohydrates as a control food) or 60 g of the fiber mix (as a drink).

Postprandial glycemic response will be assessed by changes in blood glucose levels, to be monitored using a continuous glucose monitoring system (FreeStyle Pro). A sensor will be placed on the participant's arm and will stay on until the end of the study.

Participants will provide photos of all the food and drink and a brief description of what they have consumed throughout the 2-week study.

ELIGIBILITY:
Inclusion Criteria

* Aged between 18 and 65 years
* Understand and be able to follow written and oral instructions in English
* Provide written informed consent

Exclusion Criteria

* Receiving insulin for diabetes treatment
* Receiving injectable prescription medicine
* Self-reported allergy or intolerance to any ingredients in the test food
* Any conditions deemed by the investigators that would prevent participation in the study, e.g. participation in past or active clinical research that may interfere with study outcomes, at the discretion of the investigators
* Any conditions deemed by the investigators that would compromise the individual's ability to complete the study, e.g. serious psychiatric conditions, at the discretion of the investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Postprandial glycemic response | The system will measure circulating blood glucose concentrations every 15 min continuously over 14 days. The data collected immediately prior to and up to 3 h after consuming the test food will be used to assess postprandial glycemic response
  Circulating blood glucose concentration will be measured using a continuous glucose monitoring system (FreeStyle Libre Pro, Abbott Diabetes Care)

CONTACTS AND LOCATIONS:
Overall Officials: Liping Zhao, PhD, Principal Investigator — Rutgers University
Locations (1):
- Institute for Food, Nutrition & Health, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT03334643/Prot_SAP_000.pdf